CLINICAL TRIAL: NCT03817970
Title: Drug Disposition and Nephrotoxicity
Brief Title: Cisplatin Disposition and Kidney Injury
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); Rutgers University (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-1752.cc; R01GM123330 (NIH)
Record Dates: First submitted 2018-11-27; First posted 2019-01-28 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Nephrotoxicity
Keywords: Nephrotoxicity; Cisplatin; Kidney Injury; anti-emetics
MeSH Terms: interventions — Granisetron; Ondansetron; Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Granisetron (Experimental): Participants randomized to an antiemetic regimen containing granisetron 2 mg oral or IV and evaluated for cisplatin toxicity after the first dose of cisplatin.
  Interventions: Drug: Granisetron
- Ondansetron (Experimental): Participants randomized to an antiemetic regimen containing ondansetron 8 mg oral or IV and evaluated for cisplatin toxicity after the first dose of cisplatin.
  Interventions: Drug: Ondansetron
- Palonosetron (Experimental): Participants randomized to an antiemetic regimen containing palonosetron 0.25 mg IV and evaluated for cisplatin toxicity after the first dose of cisplatin.
  Interventions: Drug: Palonosetron

INTERVENTIONS:
Drug: Granisetron — An antiemetic regimen containing granisetron 2 mg oral or IV.
  Other Names: Kytril
  Arms: Granisetron
Drug: Ondansetron — An antiemetic regimen containing ondansetron 8 mg oral or IV.
  Other Names: Zofran
  Arms: Ondansetron
Drug: Palonosetron — An antiemetic regimen containing palonosetron 0.25 mg IV.
  Other Names: Aloxi
  Arms: Palonosetron

SUMMARY:
This study is being done to determine 1) whether drugs to treat cisplatin-related nausea can influence harm to the kidneys, 2) whether cisplatin levels in the body can influence the risk of harm to the kidneys, and 3) whether a person's genetic make-up can increase or decrease the likelihood of kidney injury due to cisplatin therapy.

DETAILED DESCRIPTION:
Cisplatin (cis-diamminedichloroplatinum, Platinol®) is commonly utilized in chemotherapy regimens for the treatment of solid cancers including lung, head and neck, and cervix. Its main mechanism of action is through binding of DNA to form cross-links, leading to arrest of DNA synthesis and replication. A major adverse consequence of cisplatin therapy is acute kidney injury (AKI). It is reported that between 30 and 38 percent of patients develop signs of nephrotoxicity (toxicity in the kidneys) after a single cisplatin dose, despite strategies such as hydration to limit renal exposure. This is problematic for patients as kidney injury can delay further treatment and limit the total number of chemotherapy cycles received, thereby reducing the overall efficacy of cisplatin-containing regimens. Furthermore, it is apparent that cisplatin will remain a central component to the treatment of solid tumors in the foreseeable future. New approaches to identify patients at risk of acute kidney injury (AKI) and prevent its development and progression are urgently needed. Cisplatin causes nausea and vomiting, which requires treatment with 5-HT3 antagonists (5-HT3A) to control. Associations between the clinical use of the 5-HT3A antiemetic drugs and the risk of cisplatin AKI have recently been discovered. This study will interrogate relationships between 5-HT3A drugs (granisetron, ondansetron, and palonosetron) and cisplatin AKI.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient prescribed cisplatin at a dose of >25mg/m^2
* Age 18-80 years
* Hemoglobin >/=9 g/dl
* No consumption of grapefruit juice or alcohol within 7 days
* No history of alcohol consumption of >14 drinks/week
* No history of organ transplantation or kidney dialysis
* Willingness to comply with study
* Not pregnant or lactating
* No changes in chronic medications within 2 weeks
* Estimated glomerular filtration rate (eGFR) > 60 ml/min^2
* Normal liver function (ALT and AST <2x ULN)

Exclusion Criteria:

* Diagnosis of kidney cancer
* Previous exposure to platinum-based chemotherapy with the exception of one previous dose as part of the current course
* Herbal supplement use beyond marijuana
* Exposure to other known nephrotoxins (including contrast agents) within the previous 2 weeks
* Severe gastrointestinal disease with fluid losses
* Diagnosis of a rapidly progressive glomerulonephritis
* Allergy or contraindication to 5-HT3 Antagonists

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Kidney Injury with Cisplatin and 5-HT3 Antagonist Antiemetic Regimen as Assessed by a 1.5 fold increase in a Biomarker Panel | 3 days
  The effects of 5-HT3 antagonist antiemetic drugs on cisplatin kidney injury as indicated by a 1.5 fold increase in the urinary biomarker panel values at 3 days after treatment
The Effects of 5-HT3 Antagonist Antiemetic Drugs on Cisplatin Secretion | 3 days
  The changes to cisplatin secretion in the urine (as an early biomarker for the detection of kidney injury) as indicated by a 6 mg difference between 5-HT3 Antagonist Antiemetic Drugs at 3 days after treatment

SECONDARY OUTCOMES:
Targeted Genetic Polymorphisms are Associated with Risk of Kidney Injury Due to Cisplatin and 5-HT3 Antagonist Antiemetic Regimen as Assessed by a 1.5 fold increase in a Biomarker Panel | 3 days
  The influence of targeted genetic polymorphisms on risk of kidney injury due to cisplatin and 5-HT3 Antagonist Antiemetic Drugs as indicated by a 1.5 fold increase in a urinary biomarker panel values at 3 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Joy, PharmD, PhD, Principal Investigator — University of Colorado, Denver; Edgar Jaimes, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - UCHealth-Metro Denver, Denver, Colorado
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No